CLINICAL TRIAL: NCT05259839
Title: A Dose Escalation and Expansion Study of Etentamig (ABBV-383) in Combination With Anti-Cancer Regimens for the Treatment of Patients With Newly Diagnosed or Relapsed/Refractory Multiple Myeloma
Brief Title: A Study to Assess Adverse Events and Change in Disease Activity of Intravenously (IV) Infused Etentamig (ABBV-383) in Combination With Anti-Cancer Regimens for the Treatment of Adult Participants With Relapsed/Refractory Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M22-947; 2023-506871-88-00 (Other: EU CT)
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; Pomalidomide; Dexamethasone; Lenalidomide; Daratumumab; Nirogacestat; Etentamig; ABBV-383; Cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms | interventions — Dexamethasone; Lenalidomide; pomalidomide; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part 1: Arm A (Etentamig with Pomalidomide and Dexamethasone) (Experimental): Participants with relapsed or refractory (R/R) multiple myeloma (MM) who meet the criteria outline in the protocol will receive etentamig with Pomalidomide and Dexamethasone.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Pomalidomide
- Part 1: Arm B (Etentamig with Lenalidomide and Dexamethasone) (Experimental): Participants with R/R MM who meet the criteria outline in the protocol will receive etentamig with Lenalidomide and Dexamethasone.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Lenalidomide
- Part 1: Arm C (Etentamig with Daratumumab and Dexamethasone) (Experimental): Participants with R/R MM who meet the criteria outline in the protocol will receive etentamig with Daratumumab and Dexamethasone.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Daratumumab
- Part 2: Arm E (Etentamig with Pomalidomide and Dexamethasone) (Experimental): Participants with R/R MM who meet the criteria outline in the protocol will receive etentamig with Pomalidomide and Dexamethasone, after 1-3 prior lines of therapy.
  Interventions: Drug: Etentamig; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Etentamig — Intravenous (IV) Infusion
  Other Names: ABBV-383
Drug: Dexamethasone — Oral; Tablet or IV Infusion
Drug: Lenalidomide — Oral; Capsule
  Arms: Part 1: Arm B (Etentamig with Lenalidomide and Dexamethasone)
Drug: Pomalidomide — Oral; Capsule
  Arms: Part 1: Arm A (Etentamig with Pomalidomide and Dexamethasone); Part 2: Arm E (Etentamig with Pomalidomide and Dexamethasone)
Drug: Daratumumab — Subcutaneous Injection (SC)
  Arms: Part 1: Arm C (Etentamig with Daratumumab and Dexamethasone)

SUMMARY:
Multiple myeloma (MM) is a plasma cell disease characterized by the growth of clonal plasma cells in the bone marrow. The purpose of this study is to assess the safety and toxicity of etentamig (ABBV-383) when co-administered with pomalidomide-dexamethasone (Pd), lenalidomide-dexamethasone (Rd), or daratumumab-dexamethasone (Dd), in adult participants with relapsed/refractory (R/R) multiple myeloma (MM). Adverse events and change in disease activity will be assessed.

Etentamig is an investigational drug being developed for the treatment of R/R MM. Study doctors put the participants in groups called treatment arms. Etentamig co-administered with Pd, Rd, or Dd, will be explored. Each treatment arm receives a different treatment combination depending on stage of the study and eligibility. This study will include a dose escalation phase to determine the best dose of etentamig, followed by a dose expansion phase to confirm the dose. Approximately 320 adult participants with R/R MM will be enrolled in the study in approximately 48 sites worldwide.

Participants will receive intravenous (IV) etentamig co-administered with oral/IV Pd, oral/IV Rd, or oral/IV/subcutaneous (SC) Dd in 28-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, questionnaires and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance of <= 2.
* Must have confirmed diagnosis of Relapsed/Refractory (R/R) Multiple Myeloma (MM) with documented evidence of progression during or after the participant's last treatment regimen based on the investigator's determination of the International Myeloma Working Group (IMWG) criteria.
* Must have measurable disease as determined by central lab as outlined in the protocol.
* Must be naïve to treatment with Etentamig.
* Must have never received BCMA-targeted therapy. Participants who have received targeted therapy against non-BCMA targets will not be excluded.
* Arms A, B and C: Participant has received at least 3 prior lines of MM treatment.
* Arm E: Participant has received 1-3 prior lines of MM treatment.

Exclusion Criteria:

* Received a peripheral autologous stem cell transplant (SCT) within 12 weeks, or an allogeneic SCT within 1 year of the first dose of study treatment.
* Unresolved adverse event (AE)s >= Grade 2 (National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) from prior anticancer therapy.
* Has any of the following conditions:

  * Nonsecretory Multiple Myeloma (MM).
  * Active Plasma cell leukemia i.e., either 20% of peripheral white blood cells or > 2.0 × 10^9L circulating plasma cells by standard differential.
  * Waldenstrom's macroglobulinemia.
  * Light chain amyloidosis.
  * Polyneuropathy, organomegaly, endocrinopathy, monoclonal protein and skin changes (POEMS) syndrome.
  * Major surgery within 4 weeks prior to first dose or planned study participation.
  * Acute infections within 14 days prior to first dose of study requiring therapy (antibiotic, antifungal or antiviral).
  * Uncontrolled diabetes or hypertension within 14 days prior to first dose.
  * Peripheral neuropathy >= Grade 3 or >= Grade 2 with pain within 2 weeks prior to first dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2033-09 (Estimated); Study Completion 2033-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose Limiting Toxicities (DLT) of Etentamig | Up to approximately 28 Days
  DLT events as described in the protocol will be assessed.
Number of Participants with Adverse Events (AEs) | Up to Approximately 3 Years
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Up to Approximately 3 Years
  ORR is defined as partial response (PR) + very good partial response (VGPR) + complete remission (CR) + stringent complete response (sCR); proportion of participants who achieved a PR or better.
Progression-Free Survival (PFS) | Up to Approximately 3 Years
  PFS is defined as the number of days from the date of first dose to the date of earliest disease progression or death.
Duration of Response (DOR) | Up to Approximately 3 Years
  DOR will be defined as the number of days from the date of first response (sCR, CR, VGPR, or PR) to the earliest recurrence, progressive disease, or death, whatever occurs first.
Time-to-Progression (TTP) | Up to Approximately 3 Years
  TTP is defined as the number of days from the date of first dose to the date of earliest disease progression.
Percentage of Participants with Minimal Residual Diseas (MRD) Negativity by Next-Generation Sequencing (NGS) | Up to Approximately 3 Years
  MRD negative status (threshold as assessed by NGS Adaptive Clonoseq) with >= CR (per International Myeloma Working Group [IMWG] response criteria) prior to the initiation of new myeloma therapy.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (49):
- United States (15):
  - University of Arkansas for Medical Sciences /ID# 243096, Little Rock, Arkansas
  - Sylvester Comprehensive Cancer Center /ID# 243673, Miami, Florida
  - Moffitt Cancer Center /ID# 243437, Tampa, Florida
  - University of Maryland, Baltimore /ID# 243679, Baltimore, Maryland
  - Dana-Farber Cancer Institute /ID# 249529, Boston, Massachusetts
  - University of Massachusetts - Worcester /ID# 243977, Worcester, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 243438, Ann Arbor, Michigan
  - The Valley Hospital /ID# 243829, Paramus, New Jersey
  - Rutenberg Cancer Center /ID# 244647, New York, New York
  - Memorial Sloan Kettering Cancer Center /ID# 244656, New York, New York
  - Atrium Health Levine Cancer Institute /ID# 242851, Charlotte, North Carolina
  - University of Texas Southwestern Medical Center /ID# 243273, Dallas, Texas
  - Huntsman Cancer Institute /ID# 242872, Salt Lake City, Utah
  - University of Washington /ID# 243172, Seattle, Washington
  - Froedtert Memorial Lutheran Hospital /ID# 242654, Milwaukee, Wisconsin
- Australia (7):
  - St George Hospital /ID# 243740, Kogarah, New South Wales
  - Calvary Mater Newcastle /ID# 243730, Waratah, New South Wales
  - Monash Health - Monash Medical Centre /ID# 244403, Clayton, Victoria
  - St Vincent's Hospital Melbourne /ID# 256879, Fitzroy Melbourne, Victoria
  - Peter MacCallum Cancer Ctr /ID# 256880, Melbourne, Victoria
  - Epworth Healthcare /ID# 243734, Richmond, Victoria
  - Fiona Stanley Hospital /ID# 244753, Murdoch, Western Australia
- Germany (5):
  - Universitaetsklinikum Tuebingen /ID# 242815, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Wuerzburg /ID# 242826, Würzburg, Bavaria
  - Universitaetsklinikum Essen /ID# 242819, Essen
  - Universitaetsklinikum Hamburg-Eppendorf /ID# 243141, Hamburg
  - Universitaetsklinikum Regensburg /ID# 242837, Regensburg
- Italy (5):
  - IRCCS Ospedale San Raffaele /ID# 242583, Milan, Milano
  - Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST - IRCCS /ID# 242584, Meldola, Reggio Emilia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Universita Cattolica /ID# 242582, Rome, Roma
  - IRCCS AOU di Bologna Policlinico Sant Orsola Malpighi /ID# 242581, Bologna
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico /ID# 244057, Milan
- Japan (6):
  - Nagoya City University Hospital /ID# 249094, Nagoya, Aichi-ken
  - National Cancer Center Hospital East /ID# 245889, Kashiwa-shi, Chiba
  - Hokkaido University Hospital /ID# 245966, Sapporo, Hokkaido
  - Kanazawa University Hospital /ID# 246812, Kanazawa, Ishikawa-ken
  - Okayama Medical Center /ID# 245882, Okayama, Okayama-ken
  - Yamagata University Hospital /ID# 245888, Yamagata, Yamagata
- Poland (4):
  - Szpital Wojewodzki w Opolu sp. z o.o. /ID# 243954, Opole, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny We Wrocławiu /ID# 243246, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie /ID# 243500, Lublin, Lublin Voivodeship
  - Uniwersyteckie Centrum Kliniczne /ID# 243249, Gdansk, Pomeranian Voivodeship
- Spain (7):
  - Hospital Duran i Reynals /ID# 242979, L'Hospitalet de Llobregat, Barcelona
  - Clinica Universidad de Navarra - Pamplona /ID# 242977, Pamplona, Navarre
  - Hospital Universitario Vall de Hebron /ID# 242976, Barcelona
  - Hospital Clinic de Barcelona /ID# 242978, Barcelona
  - CLINICA UNIVERSIDAD DE NAVARRA-Madrid /ID# 244145, Madrid
  - Hospital Universitario 12 de Octubre /ID# 242975, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 242974, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-947